CLINICAL TRIAL: NCT01018537
Title: NARCOMS Global Multiple Sclerosis Registry: A Long-Term Study to Facilitate Research in Multiple Sclerosis
Brief Title: NARCOMS Registry: A Multiple Sclerosis Registry
Acronym: NARCOMS
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Consortium of Multiple Sclerosis Centers (Other)
Responsible Party: Principal Investigator, Amber Salter, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: 20081794
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; NARCOMS; Patient Registry; Registry
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
This project is based on the idea that we can learn about the complexities of MS by following disease and treatment patterns in a large group of people over several years. The information gathered is used for research only. Results are presented in summary form only. All details submitted by registry participants is strictly confidential.

To participate in NARCOMS complete the baseline enrollment survey online through www.narcoms.org (or directly using the following link: https://redcap.link/py2rnyyn) or you can request a mail-in survey be sent to you by emailing MSregistry@narcoms.org. You will be asked to update your information, online or by mail, twice a year. Each update survey typically takes less than 20 minutes to complete.

There is no cost to participate. For your participation you are offered a free subscription to the NARCOMS quarterly magazine, NARCOMS Now. NARCOMS Now provides a reliable source of information about the latest in MS research and disease management. You can stop participating in the registry at any time.

You may also receive additional surveys or information on clinical trials. You are not obligated to participate and these additional studies will always come directly from NARCOMS. Your contact information will not be shared or sold to other parties.

DETAILED DESCRIPTION:
The data coordinating center, located at the University of Texas Southwestern Medical Center, maintains NARCOMS, the worlds largest voluntary, patient driven MS registry. The registry involves personnel from at least three other sites in the US and Canada (Cleveland Clinic Foundation, University of Alabama at Birmingham, and the Dalhousie University in Canada). Over the past 30 years more than 42,000 people with MS across the U.S., Canada and over 50 other countries, including over 4,000 Veterans, have participated in the registry by submitting their health-related data by mail or online. Registry data have been featured in over 100 peer-reviewed journal articles, scientific posters and presentations. These reports have provided information to guide new research. They also provide evidence supporting the approval of new drugs in the fight against MS.

The North American Research Committee on Multiple Sclerosis (NARCOMS) is supported in part by the Consortium of Multiple Sclerosis Centers (CMSC), a not-for-profit professional organization for multiple sclerosis (MS) healthcare providers and researchers involving 198 participating centers of the MS treatment and research community.

ELIGIBILITY:
Inclusion Criteria:

* Any individual who has been diagnosed with multiple sclerosis or clinically isolated syndrome
* Must be at least 18 years of age

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have been diagnosed with multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 1996-01; Primary Completion 2050-12 (Estimated); Study Completion 2050-12 (Estimated)

PRIMARY OUTCOMES:
Disease progression over time of follow up | up to 15 years
  Disease Progression measured using the Patient Determined Disease Steps

SECONDARY OUTCOMES:
Contributing factors to change in MS disease status | up to 15 years
  Factors include, but not limited to, demographics, lifestyle and clinical characteristics

OTHER OUTCOMES:
Medication usage in multiple sclerosis | up to 15 years
  Disease modifying therapy use is collected from participants

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Fox, M.D., Study Director — Mellen Center for MS / Cleveland Clinic; Amber Salter, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center; Gary R Cutter, Ph.D., Study Director — University of Alabama at Birmingham; Ruth Ann Marrie, M.D., Ph.D., Study Director — Dalhousie University
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Mahajan ST, Patel PB, Marrie RA. Under treatment of overactive bladder symptoms in patients with multiple sclerosis: an ancillary analysis of the NARCOMS Patient Registry. J Urol. 2010 Apr;183(4):1432-7. doi: 10.1016/j.juro.2009.12.029. Epub 2010 Feb 20. PMID 20171697
- [Background] Buchanan RJ, Chakravorty BJ, Tyry T, Hatcher W, Vollmer T. Age-related comparisons of people with multiple sclerosis: demographic, disease, and treatment characteristics. NeuroRehabilitation. 2009;25(4):271-8. doi: 10.3233/NRE-2009-0525. PMID 20037220
- [Background] Marrie RA, Cutter G, Tyry T, Vollmer T. A cross-sectional study of bone health in multiple sclerosis. Neurology. 2009 Oct 27;73(17):1394-8. doi: 10.1212/WNL.0b013e3181beece8. PMID 19858462
- [Background] Hadjimichael O, Vollmer T, Oleen-Burkey M; North American Research Committee on Multiple Sclerosis. Fatigue characteristics in multiple sclerosis: the North American Research Committee on Multiple Sclerosis (NARCOMS) survey. Health Qual Life Outcomes. 2008 Nov 14;6:100. doi: 10.1186/1477-7525-6-100. PMID 19014588
- [Background] Marrie RA, Cutter G, Tyry T, Campagnolo D, Vollmer T. Smoking status over two years in patients with multiple sclerosis. Neuroepidemiology. 2009;32(1):72-9. doi: 10.1159/000170910. Epub 2008 Nov 12. PMID 19001800
- [Background] Marrie R, Horwitz R, Cutter G, Tyry T, Campagnolo D, Vollmer T. High frequency of adverse health behaviors in multiple sclerosis. Mult Scler. 2009 Jan;15(1):105-13. doi: 10.1177/1352458508096680. Epub 2008 Oct 9. PMID 18845651
- [Background] Marrie R, Horwitz R, Cutter G, Tyry T, Campagnolo D, Vollmer T. Comorbidity, socioeconomic status and multiple sclerosis. Mult Scler. 2008 Sep;14(8):1091-8. doi: 10.1177/1352458508092263. PMID 18728060
- [Background] Julian LJ, Vella L, Vollmer T, Hadjimichael O, Mohr DC. Employment in multiple sclerosis. Exiting and re-entering the work force. J Neurol. 2008 Sep;255(9):1354-60. doi: 10.1007/s00415-008-0910-y. Epub 2008 Jul 17. PMID 18677639
- [Background] Marrie RA, Cutter G, Tyry T, Vollmer T, Campagnolo D. Disparities in the management of multiple sclerosis-related bladder symptoms. Neurology. 2007 Jun 5;68(23):1971-8. doi: 10.1212/01.wnl.0000264416.53077.8b. PMID 17548546
- [Background] Marrie RA, Cutter G, Tyry T, Campagnolo D, Vollmer T. Validation of the NARCOMS registry: diagnosis. Mult Scler. 2007 Jul;13(6):770-5. doi: 10.1177/1352458506075031. Epub 2007 Mar 15. PMID 17525097
- [Background] Hadjimichael O, Kerns RD, Rizzo MA, Cutter G, Vollmer T. Persistent pain and uncomfortable sensations in persons with multiple sclerosis. Pain. 2007 Jan;127(1-2):35-41. doi: 10.1016/j.pain.2006.07.015. Epub 2006 Sep 1. PMID 16949751
- [Background] Kobelt G, Berg J, Atherly D, Hadjimichael O. Costs and quality of life in multiple sclerosis: a cross-sectional study in the United States. Neurology. 2006 Jun 13;66(11):1696-702. doi: 10.1212/01.wnl.0000218309.01322.5c. PMID 16769943
- [Background] Marrie RA, Cutter G, Tyry T, Vollmer T, Campagnolo D. Does multiple sclerosis-associated disability differ between races? Neurology. 2006 Apr 25;66(8):1235-40. doi: 10.1212/01.wnl.0000208505.81912.82. PMID 16636241
- [Background] Marrie RA, Cutter G, Tyry T, Hadjimichael O, Campagnolo D, Vollmer T. Changes in the ascertainment of multiple sclerosis. Neurology. 2005 Oct 11;65(7):1066-70. doi: 10.1212/01.wnl.0000178891.20579.64. PMID 16217060
- [Background] Marrie RA, Cutter G, Tyry T, Hadjimichael O, Campagnolo D, Vollmer T. Validation of the NARCOMS registry: fatigue assessment. Mult Scler. 2005 Oct;11(5):583-4. doi: 10.1191/1352458505ms1216oa. PMID 16193897
- [Background] Marrie RA, Cutter G, Tyry T, Hadjimichael O, Vollmer T. Validation of the NARCOMS Registry: pain assessment. Mult Scler. 2005 Jun;11(3):338-42. doi: 10.1191/1352458505ms1167oa. PMID 15957517
- [Background] Lo AC, Hadjimichael O, Vollmer TL. Treatment patterns of multiple sclerosis patients: a comparison of veterans and non-veterans using the NARCOMS registry. Mult Scler. 2005 Feb;11(1):33-40. doi: 10.1191/1352458505ms1136oa. PMID 15732264
- [Background] Rizzo MA, Hadjimichael OC, Preiningerova J, Vollmer TL. Prevalence and treatment of spasticity reported by multiple sclerosis patients. Mult Scler. 2004 Oct;10(5):589-95. doi: 10.1191/1352458504ms1085oa. PMID 15471378
- [Background] Marrie RA, Hadjimichael O, Vollmer T. Predictors of alternative medicine use by multiple sclerosis patients. Mult Scler. 2003 Oct;9(5):461-6. doi: 10.1191/1352458503ms953oa. PMID 14582770
- [Background] Buchanan RJ, Radin D, Chakravorty BJ, Tyry T. Informal care giving to more disabled people with multiple sclerosis. Disabil Rehabil. 2009;31(15):1244-56. doi: 10.1080/09638280802532779. PMID 19802928
- [Background] Buchanan R, Radin D, Chakravorty BJ, Tyry T. Perceptions of informal care givers: health and support services provided to people with multiple sclerosis. Disabil Rehabil. 2010;32(6):500-10. doi: 10.3109/09638280903171485. PMID 19852704
- [Background] Finlayson M, Cho C. A descriptive profile of caregivers of older adults with MS and the assistance they provide. Disabil Rehabil. 2008;30(24):1848-57. doi: 10.1080/09638280701707324. PMID 18608376
- [Background] Fraser C, Hadjimichael O, Vollmer T. Predictors of adherence to glatiramer acetate therapy in individuals with self-reported progressive forms of multiple sclerosis. J Neurosci Nurs. 2003 Jun;35(3):163-70. doi: 10.1097/01376517-200306000-00006. PMID 12830664
- [Background] Fraser C, Morgante L, Hadjimichael O, Vollmer T. A prospective study of adherence to glatiramer acetate in individuals with multiple sclerosis. J Neurosci Nurs. 2004 Jun;36(3):120-9. doi: 10.1097/01376517-200406000-00002. PMID 15233411
- [Background] Marrie RA, Horwitz R, Cutter G, Tyry T, Campagnolo D, Vollmer T. Comorbidity delays diagnosis and increases disability at diagnosis in MS. Neurology. 2009 Jan 13;72(2):117-24. doi: 10.1212/01.wnl.0000333252.78173.5f. Epub 2008 Oct 29. PMID 18971448
- [Background] Marrie RA, Rudick R, Horwitz R, Cutter G, Tyry T, Campagnolo D, Vollmer T. Vascular comorbidity is associated with more rapid disability progression in multiple sclerosis. Neurology. 2010 Mar 30;74(13):1041-7. doi: 10.1212/WNL.0b013e3181d6b125. PMID 20350978
- [Background] Buchanan RJ, Minden SL, Chakravorty BJ, Hatcher W, Tyry T, Vollmer T. A pilot study of young adults with multiple sclerosis: demographic, disease, treatment, and psychosocial characteristics. Disabil Health J. 2010 Oct;3(4):262-70. doi: 10.1016/j.dhjo.2009.09.003. Epub 2009 Nov 26. PMID 21122795
- [Background] Marrie RA, Horwitz RI, Cutter G, Tyry T, Vollmer T. Association between comorbidity and clinical characteristics of MS. Acta Neurol Scand. 2011 Aug;124(2):135-41. doi: 10.1111/j.1600-0404.2010.01436.x. Epub 2010 Sep 29. PMID 20880264
- [Background] Salter AR, Cutter GR, Tyry T, Marrie RA, Vollmer T. Impact of loss of mobility on instrumental activities of daily living and socioeconomic status in patients with MS. Curr Med Res Opin. 2010 Feb;26(2):493-500. doi: 10.1185/03007990903500649. PMID 20014979
- [Background] Buchanan RJ, Zuniga MA, Carrillo-Zuniga G, Chakravorty BJ, Tyry T, Moreau RL, Huang C, Vollmer T. Comparisons of Latinos, African Americans, and Caucasians with multiple sclerosis. Ethn Dis. 2010 Autumn;20(4):451-7. PMID 21305836
- [Background] Marrie RA, Horwitz R, Cutter G, Tyry T. Cumulative impact of comorbidity on quality of life in MS. Acta Neurol Scand. 2012 Mar;125(3):180-6. doi: 10.1111/j.1600-0404.2011.01526.x. Epub 2011 May 26. PMID 21615355
- [Background] Marrie RA, Horwitz RI, Cutter G, Tyry T, Vollmer T. Smokers with multiple sclerosis are more likely to report comorbid autoimmune diseases. Neuroepidemiology. 2011;36(2):85-90. doi: 10.1159/000323948. Epub 2011 Feb 1. PMID 21282965
- [Background] Cutter GR, Zimmerman J, Salter AR, Knappertz V, Suarez G, Waterbor J, Howard VJ, Marrie RA. Causes of death among persons with multiple sclerosis. Mult Scler Relat Disord. 2015 Sep;4(5):484-490. doi: 10.1016/j.msard.2015.07.008. Epub 2015 Jul 18. PMID 26346799
- [Background] Bethoux F, Marrie RA. A Cross-Sectional Study of the Impact of Spasticity on Daily Activities in Multiple Sclerosis. Patient. 2016 Dec;9(6):537-546. doi: 10.1007/s40271-016-0173-0. PMID 27154536
- [Background] Wang G, Marrie RA, Salter AR, Fox R, Cofield SS, Tyry T, Cutter GR. Health insurance affects the use of disease-modifying therapy in multiple sclerosis. Neurology. 2016 Jul 26;87(4):365-74. doi: 10.1212/WNL.0000000000002887. Epub 2016 Jun 29. PMID 27358338
- [Background] Salter A, Tyry T, Wang G, Fox RJ, Cutter G, Marrie RA. Examining the joint effect of disability, health behaviors, and comorbidity on mortality in MS. Neurol Clin Pract. 2016 Oct;6(5):397-408. doi: 10.1212/CPJ.0000000000000269. PMID 27847682
- [Background] Salter A, Thomas N, Tyry T, Cutter G, Marrie RA. Employment and absenteeism in working-age persons with multiple sclerosis. J Med Econ. 2017 May;20(5):493-502. doi: 10.1080/13696998.2016.1277229. Epub 2017 Jan 25. PMID 28035846
- [Background] Reider N, Salter AR, Cutter GR, Tyry T, Marrie RA. Potentially Modifiable Factors Associated With Physical Activity in Individuals With Multiple Sclerosis. Res Nurs Health. 2017 Apr;40(2):143-152. doi: 10.1002/nur.21783. Epub 2017 Feb 6. PMID 28165143
- [Background] Marrie RA, Salter A, Tyry T, Cutter GR, Cofield S, Fox RJ. High hypothetical interest in physician-assisted death in multiple sclerosis. Neurology. 2017 Apr 18;88(16):1528-1534. doi: 10.1212/WNL.0000000000003831. Epub 2017 Mar 15. PMID 28298551
- [Background] Marrie RA, Cutter GR, Tyry T, Cofield SS, Fox R, Salter A. Upper limb impairment is associated with use of assistive devices and unemployment in multiple sclerosis. Mult Scler Relat Disord. 2017 Apr;13:87-92. doi: 10.1016/j.msard.2017.02.013. Epub 2017 Feb 20. PMID 28427709
- [Background] Salter A, Thomas NP, Tyry T, Cutter GR, Marrie RA. A contemporary profile of primary progressive multiple sclerosis participants from the NARCOMS Registry. Mult Scler. 2018 Jun;24(7):951-962. doi: 10.1177/1352458517711274. Epub 2017 May 19. PMID 28524746
- [Background] Marrie RA, Sharma M, Cutter GR, Fox RJ, Salter A. Perspectives of People With Multiple Sclerosis Regarding Data Linkage and Sharing. Neurology. 2025 May 13;104(9):e213587. doi: 10.1212/WNL.0000000000213587. Epub 2025 Apr 8. PMID 40198867
- [Background] Salter A, Lancia S, Sharma M, Cutter GR, Fox RJ, Marrie RA. Infection, Relapses, and Pseudo-Relapses in Individuals With Multiple Sclerosis. Neurol Clin Pract. 2025 Aug;15(4):e200493. doi: 10.1212/CPJ.0000000000200493. Epub 2025 Jun 4. PMID 40510870
- [Background] Salter A, Lancia S, Cutter GR, Fox RJ, Marrie RA. Effects of COVID-19 Infection on Symptom Severity and Disability in Multiple Sclerosis. Neurology. 2025 Jan 28;104(2):e210149. doi: 10.1212/WNL.0000000000210149. Epub 2024 Dec 23. PMID 39715473
- [Background] O'Mahony J, Salter A, Ciftci-Kavaklioglu B, Fox RJ, Cutter GR, Marrie RA. Physical and Mental Health-Related Quality of Life Trajectories Among People With Multiple Sclerosis. Neurology. 2022 Oct 3;99(14):e1538-e1548. doi: 10.1212/WNL.0000000000200931. PMID 35948450
- [Background] Marrie RA, Cutter GR, Fox RJ, Vollmer T, Tyry T, Salter A. NARCOMS and Other Registries in Multiple Sclerosis: Issues and Insights. Int J MS Care. 2021 Nov-Dec;23(6):276-284. doi: 10.7224/1537-2073.2020-133. Epub 2021 Dec 29. PMID 35035299
- See also: NARCOMS homepage where you can get more information or enroll in the registry. — http://www.narcoms.org
- See also: Consortium of Multiple Sclerosis Centers (CMSC) homepage — https://mscare.org
- See also: NARCOMS PubMed Bibliography — https://www.ncbi.nlm.nih.gov/myncbi/1pqyrIe3kbgQ7/bibliography/public/